CLINICAL TRIAL: NCT06182644
Title: Head-to-head Comparison of Positron Nuclide Radio-labeled FAPI and 18F-FDG PET/CT in Patients With Malignant Tumors
Acronym: FAPI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Guangdong
Record Dates: First submitted 2023-12-08; First posted 2023-12-27 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-12

CONDITIONS: Renal Cell Carcinoma; Gastric Cancer; Hepatocellular Carcinoma; Signet Ring Cell Carcinoma; Mucinous Adenocarcinoma; Colorectal Cancer
Keywords: FAPI PET/CT; FDG PET/CT
MeSH Terms: conditions — Carcinoma, Renal Cell; Stomach Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Signet Ring Cell; Adenocarcinoma, Mucinous; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Positron-labeled FAPI PET/CT (Experimental): Imaging was performed 60 minutes after injection of 5mci Positron-labeled FAPI tracer
  Interventions: Diagnostic Test: FAPI PET/CT

INTERVENTIONS:
Diagnostic Test: FAPI PET/CT — The same group of patients underwent FAPI PET/CT and FDG PET/CT examinations respectively
  Other Names: FDG PET/CT examinations

SUMMARY:
The latest research has found that the use of positron-labeled FAP inhibitors for targeting FAP has achieved very good results in displaying tumor stroma, especially for tumors with poor FDG PET/CT observation, such as liver cancer, renal cancer, and gastric cancer. Although the studies were based on small sample data or case reports, they achieved significantly better results than 18F-FDG [13,15-17].

For patients who meet the inclusion and exclusion criteria, using FAPI PET/CT and FDG PET/CT imaging may have guiding significance for your treatment. If distant metastasis is found, information such as the location, size, and quantity of metastasis can be provided to provide objective imaging information for further treatment; We will promptly provide detailed information to you and your supervising physician, who will guide your personalized treatment.

The drugs used have undergone strict quality inspection, and currently, no adverse reactions have been found in multiple medical institutions both domestically and internationally. If you experience any discomfort, new changes in your condition, or any unexpected circumstances during the study period, regardless of whether it is related to the study or not, you should promptly notify your doctor or contact our research leader. He/she will make a judgment and provide appropriate medical treatment. We will provide a certain proportion of compensation for any additional visits and expenses incurred during this examination. The entire research process is under the supervision of relevant departments of Guangdong Provincial People's Hospital. If you encounter any questions during the research process, you can consult the research doctor.

DETAILED DESCRIPTION:
At the beginning of 2022, the National Cancer Center released the latest statistical data showing that the incidence rate of malignant tumors in China reached 293.91/100000, and the mortality rate reached 174.55/100000 [1]. Malignant tumors have become an important public health issue affecting the health of Chinese residents, bringing a heavy economic burden to the public health system. Different from the cancer spectrum in developed countries, digestive system tumors with poor prognosis in China, such as lung cancer, liver cancer, stomach cancer, intestinal cancer, and esophageal cancer, are at a high incidence, while those with good prognosis in European and American developed countries are at a high incidence, such as thyroid cancer, breast cancer and prostate cancer; Even the 5-year survival rate of thyroid cancer, breast cancer and prostate cancer with good prognosis still lags behind that of developed countries such as the United States [2,3]. The main reason for this is the low number of early cases, low early diagnosis rate, and non-standard clinical diagnosis and treatment of late cases. Therefore, early detection, diagnosis, staging, and intervention have become urgent issues to be addressed.

Malignant tumors often have insidious onset and overlapping symptoms; Most patients are discovered by chance, and when clinical symptoms and signs are more obvious, patients are often in the late clinical stage. Relying solely on serum tumor markers for diagnosis may result in certain false positives and false negatives [5]. Imaging examination is the preferred and non-invasive evaluation method for malignant tumors, with the advantages of being intuitive and simple. Ultrasound imaging has the advantages of non-invasive, convenient, and high accuracy in the diagnosis of superficial organs such as the thyroid, breast, and liver. However, the detection results are greatly influenced by the examiner's experience, and the repeatability is poor. Its application in staging, efficacy evaluation, and prognosis follow-up is limited. CT and MR scans can provide detailed and accurate anatomical information for identifying the location of the primary lesion, local and distant metastases, and are crucial for determining the optimal surgical plan and treatment selection [6]. However, the accuracy of anatomical imaging is limited by the size and morphology of the lesion, and small lesions are prone to misdiagnosis. In addition, some malignant tumor lesions have concealment, making them difficult to detect and diagnose.

The emergence of functional imaging devices has made real-time fusion of anatomical structures and functional/metabolic/biochemical images possible. Positron emission computed tomography/X-ray computed tomography (PET/CT) uses specific molecular probes to target tumor visualization. It can provide detailed information on the biochemical changes of tumor tissue at the cellular and molecular levels, with better sensitivity and specificity compared to traditional imaging methods, achieving the goal of accurate diagnosis [7-9]. 18F-FDG is currently the most widely used positron imaging agent in clinical practice, with good sensitivity and specificity for lung cancer. 18F-FDG is not a tumor-specific imaging agent and is susceptible to interference from patient eating and blood glucose levels; Before examination, the patient needs to have an empty stomach for at least 6 hours, and the blood sugar level needs to be lower than 11.0mmol/L, which is difficult for some diabetes patients to tolerate. The physiological uptake of brain, myocardium, intestinal mucosa, infected tissue, or inflammatory cells can lead to high uptake of 18F-FDG, resulting in a significant increase in false positive rates; In addition, some tumors, such as well-differentiated hepatocellular carcinoma, renal cell carcinoma, and signet ring cell carcinoma, have a low uptake rate of 18F-FDG and a high false negative rate. Therefore, developing new tumor-targeted molecular probes is very important [10,11].

The latest research found that in tumor tissues, especially epithelial tumors, such as ovarian cancer, gastric cancer, lung cancer, and breast cancer, the tumor matrix fibroblast membrane highly expresses fibroblast activation protein (FAP), which is a type II transmembrane serine protease [12,13]. It is worth noting that the liver, ovaries, pancreas, and stomach hardly exhibit FAP activity under normal conditions, but after carcinogenesis, the expression level of FAP is significantly increased. Therefore, based on the upregulation and selective expression of FAP after normal tissue carcinogenesis, it has been identified as a potential biomarker for tumor-associated fibroblasts [14]. In recent years, foreign scholars have achieved very good results in using positron-labeled FAP inhibitors to target FAP and display tumor stroma. Although the studies were based on small sample data or case reports, they achieved significantly better results than 18F-FDG [13,15-17]. Therefore, further multi-case and head-to-head studies with 18F-FDG are necessary for various malignant tumors.

Therefore, this study used an intra-individual control to compare the head-to-head comparison between positron-labeled fibroblast activation protein inhibitors and 18F-FDG PET/CT in detecting primary and metastatic lesions of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high clinical suspicion of malignant tumors;
2. Those who have undergone endoscopic biopsy or puncture biopsy indicating malignant tumors but have not undergone surgery or chemotherapy;
3. Previous history of malignant tumor surgery, suspected of recurrence or distant metastasis;
4. There is a willingness for puncture biopsy or surgery, and there are no contraindications for puncture biopsy or surgery, and there are no contraindications for anesthesia;
5. Sign an informed consent form and undergo a nuclear medicine examination, without any contraindications, with the ability and willingness to participate in the follow-up plan.

Exclusion Criteria:

1. Those who cannot tolerate puncture biopsy or surgical contraindications;
2. Those who have undergone radiotherapy and chemotherapy in the past 3 months;
3. Individuals who are allergic to multiple drugs or foods;
4. Those who refuse nuclear medicine examinations;
5. Those who do not agree to sign an informed consent form and are unable or willing to follow up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
SUVmax (Standardized Uptake Value max) | Within 24 hours after the patient's PET/CT scan is completed
  Manual delineation of the area of interest to measure the maximum standard uptake values of the primary lesion and each metastatic lesion

SECONDARY OUTCOMES:
Tumor-to-background ratios | Within 24 hours after the patient's PET/CT scan is completed
  Manually delineate the area of interest to measure the maximum standard uptake value (SUVmax) of the primary lesion and each metastatic lesion, as well as the average standard uptake value (SUVmean) in the liver and ascending aorta. Using the SUVmax/SUVmean ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Case Record Form and Electronic Collection and Management System
Supporting Information: Study Protocol, SAP
Time Frame: Within 2 years after the completion of the study
Access Criteria: Case Record Form and Electronic Collection and Management System
URL: https://www.gdghospital.org.cn

REFERENCES:
- [Background] Wang L, Tang G, Hu K, Liu X, Zhou W, Li H, Huang S, Han Y, Chen L, Zhong J, Wu H. Comparison of 68Ga-FAPI and 18F-FDG PET/CT in the Evaluation of Advanced Lung Cancer. Radiology. 2022 Apr;303(1):191-199. doi: 10.1148/radiol.211424. Epub 2022 Jan 4. PMID 34981976
- [Background] Pang Y, Zhao L, Luo Z, Hao B, Wu H, Lin Q, Sun L, Chen H. Comparison of 68Ga-FAPI and 18F-FDG Uptake in Gastric, Duodenal, and Colorectal Cancers. Radiology. 2021 Feb;298(2):393-402. doi: 10.1148/radiol.2020203275. Epub 2020 Dec 1. PMID 33258746